CLINICAL TRIAL: NCT00027729
Title: Phase I/II Study of MEDI-522, A Humanized Monoclonal Antibody Directed Against the Human Alpha V Beta 3 Integrin, in Patients With Irinotecan-Refractory Advanced Colorectal Cancer
Brief Title: Monoclonal Antibody Therapy in Treating Patients With Advanced Colorectal Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: 01-078; CDR0000069061 (Registry Identifier: PDQ (Physician Data Query)); MEDIMMUNE-MI-CP068; NCI-G01-2032
Record Dates: First submitted 2001-12-07; First posted 2003-01-27 (Estimated); Last update posted 2013-06-05 (Estimated); Status verified 2013-06

CONDITIONS: Colorectal Cancer
Keywords: recurrent colon cancer; recurrent rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — etaracizumab

INTERVENTIONS:
Biological: etaracizumab

SUMMARY:
RATIONALE: Monoclonal antibodies can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells.

PURPOSE: Phase I/II trial to study the effectiveness of monoclonal antibody therapy in treating patients who have advanced colorectal cancer that has not responded to irinotecan.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the recommended phase II dose of monoclonal antibody anti-anb3 integrin in patients with irinotecan-refractory advanced colorectal cancer.
* Determine the safety and tolerance of this drug in these patients.
* Determine any antitumor activity of this drug in these patients.
* Determine the objective response rate, response duration, and time to progression in patients treated with this drug.
* Determine the pharmacokinetics of this drug in these patients.

OUTLINE: This is a dose-escalation study.

Patients receive monoclonal antibody anti-anb3 integrin IV over 30 minutes once weekly on weeks 1-52 in the absence of disease progression or unacceptable toxicity. Patients with responding disease may continue therapy.

Cohort of 4-6 patients receive escalating doses of monoclonal antibody anti-anb3 integrin until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 4 or 6 patients experience dose-limiting toxicity. Once the MTD is determined, additional patients are treated at that dose in the phase II portion of the study.

Patients are followed every 3 months for 2 years.

PROJECTED ACCRUAL: A total of 4-24 patients will be accrued for phase I of this study and a total of 40 patients will be accrued for phase II of this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed advanced colorectal cancer
* Disease progression while receiving an irinotecan-containing regimen for metastatic colorectal cancer OR
* Disease recurrence within 6 months after completing an irinotecan-containing regimen in the adjuvant setting
* At least 1 measurable lesion (for phase II only)

  * At least 20 mm by x-ray, CT scan, MRI, or photograph
  * Recurrent disease after surgery or radiotherapy is considered measurable if it has been at least 4 weeks since treatment and measurable disease is outside the port of prior radiotherapy or there is evidence of disease progression within the port of prior radiotherapy
  * The following are not considered measurable:

    * Pleural effusion
    * Ascites
    * Osteoblastic lesion or evidence of disease on bone scan alone
    * Progressive irradiated lesions alone
    * Bone marrow involvement
    * Brain metastases
    * Malignant hepatomegaly by physical exam alone
    * Chemical markers (e.g., carcinoembryonic antigen)
* No known brain metastases or primary brain tumors
* No symptomatic pleural effusion or ascites requiring paracentesis
* No clinical evidence of bowel obstruction

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-1

Life expectancy:

* Not specified

Hematopoietic:

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin greater than 10.0 g/dL

Hepatic:

* Bilirubin no greater than 2.0 mg/dL
* AST/ALT no greater than 5 times upper limit of normal (ULN)
* PT/PTT less than ULN OR
* INR less than 1.12
* No hepatitis virus infection

Renal:

* Creatinine no greater than 1.5 mg/dL OR
* Creatinine clearance greater than 50 mL/min

Cardiovascular:

* No prior myocardial infarction
* No angina
* No uncontrolled hypertension (systolic blood pressure greater than 150 mm Hg)
* No prior cerebrovascular accident or transient ischemic attack

Pulmonary:

* No respiratory insufficiency requiring oxygen treatment
* No lymphangitic involvement of lungs

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception for 30 days before, during, and for 30 days after study
* Thyroxine and thyroid-stimulating hormone normal
* No hematemesis, melena, hematochezia, or gross hematuria
* No prior significant adverse reaction to a humanized monoclonal antibody
* No known HIV infection
* No active infection requiring systemic anti-infective therapy
* No other medical or psychological condition or behavior, including substance dependence or abuse, that would preclude study
* No other malignancy within the past 5 years except basal cell skin cancer or completely excised carcinoma in situ of the cervix

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Prior immunotherapy with approved agents allowed
* No prior monoclonal antibody anti-anb3 integrin or its precursor (MEDI-523)
* No other concurrent immunotherapy

Chemotherapy:

* See Disease Characteristics
* At least 4 weeks since prior chemotherapy
* No concurrent palliative chemotherapy

Endocrine therapy:

* No concurrent hormonal therapy

Radiotherapy:

* See Disease Characteristics
* At least 4 weeks since prior radiotherapy

Surgery:

* See Disease Characteristics
* At least 4 weeks since prior surgery and surgical wounds must have healed

Other:

* Recovered from all prior therapy
* At least 4 weeks since prior investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-06; Primary Completion 2004-11 (Actual); Study Completion 2004-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leonard B. Saltz, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States